CLINICAL TRIAL: NCT06255899
Title: Does Adding Individualized Feedback on Movement Improve Effectiveness of an Injury Prevention Program in Female Lacrosse Athletes?
Brief Title: Injury Prevention for Female Lacrosse Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Sara Gombatto, Professor, San Diego State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HS-2022-0259
Record Dates: First submitted 2023-01-06; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Lower Extremity Problem
Keywords: injury prevention program; biomechanics; education; feedback; female; lacrosse; athletes

STUDY DESIGN:
Intervention Model Description: The pilot study model is a single site, 2-arm parallel quasi-experimental intervention study. After completing the baseline testing, enrolled participants will be purposively assigned (non-random) to one of two intervention groups, control (education only) or education with individualized feedback, which will be balanced based on position, playing time, and history of injury.
Masking Description: Participants, care providers, investigators and primary outcomes assessors will not be masked. Standardized procedures and scripts will be used to ensure consistency of conducting biomechanical assessments for primary outcomes in the absence of masking outcomes assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education (Active Comparator): All participants will attend an educational training session on the team's Injury Prevention Program (IPP), which will be performed prior to practices and matches throughout the season. All team members, coaching staff, and medical staff will attend the educational session. This session will be administered during the pre-season training period, will last 60-90 minutes, and include a didactic component and a practical component in which all athletes on the team will receive instruction on how to properly perform each component of the IPP program. and have an opportunity to practice performing the IPP on the field. This is an evidence-based program that will be provided to all lacrosse athletes regardless of participation in the research study.
  Interventions: Behavioral: Education Program on Injury Prevention
- Individualized Feedback + Education (Experimental): After completing the Education Program, participants assigned to the individualized feedback group will perform the IPP during a strength and conditioning session while a research team member records their performance on a laboratory video camera. The video will be analyzed to identify errors and compensations with movements and a plan for a feedback session to correct movements will be developed. The feedback session will include showing the athlete their video, identifying the error or compensation, and providing verbal, tactile, and visual feedback to correct the error or compensation. Two additional feedback sessions will be scheduled at regular intervals during the season.
  Interventions: Behavioral: Education Program on Injury Prevention; Behavioral: Individualized Feedback + Education Program on Injury Prevention

INTERVENTIONS:
Behavioral: Education Program on Injury Prevention — The didactic component of the injury prevention education program includes information on prevalence of injuries in female athletes, biomechanical risk factors for injury, and effectiveness of injury prevention programs (IPP) for mitigation of injury risk. Examples of different activities from the IPP, including proper and improper movement strategies will be provided. Athletes will be instructed as a group on how to properly perform of each activity of the IPP, and will be given an opportunity to practice. Athletes, coaches, and staff will be provided with links to written instructions and videos of proper performance for each activity. The IPP will be performed at least 3 times/week prior to practice. Coaches, staff, and athletes will be encouraged to provide supervision and feedback on performance of the IPP throughout the season.
Behavioral: Individualized Feedback + Education Program on Injury Prevention — In addition to the education program, participants in this group will receive individualized feedback on performance of the IPP. The participant will be videotaped while performing the IPP, and movement errors and compensations will be identified to provide a basis for feedback sessions to correct movement. The session will include different forms of feedback including showing the athlete their video, identifying the error or compensation, and providing verbal, tactile, and visual feedback to correct the error or compensation. Common errors and compensations, along with verbal cues and corrections, have been identified and manualized for the study. Two additional feedback sessions will be scheduled at regular intervals during the season to provide feedback on performance throughout the season. Participants in this group will be encouraged to provide peer feedback to one another.
  Arms: Individualized Feedback + Education

SUMMARY:
In this pilot study the investigators are testing whether an injury prevention program will help improve quality of movement and decrease number of injuries in collegiate women's lacrosse athletes. The primary purpose is to determine whether an injury prevention program including individualized movement instruction along with an educational program is better than an educational program alone for improving movements that can increase risk of injury and decreasing number of injuries. The investigators will recruit women's lacrosse athletes from the San Diego State University women's lacrosse team. Enrolled participants will be divided up into two groups of 10 individuals. Both groups will participate in an injury prevention educational program including a lecture component with pictures and videos, and a practice component in which athletes will be provided with group instruction on how to perform the activities and then will have an opportunity to practice all activities. In addition to the educational program, athletes in the individualized movement instruction group will be provided individualized feedback on their movements when performing activities from the injury prevention program during 3 sessions throughout the season. The primary outcomes that will be evaluated include lower body movement during a jumping and balance task as measured using a 3D motion capture system. The investigators hypothesize that participants who receive the individualized feedback in addition to the education program will display greater improvements in movements that increase injury risk when compare to the education only intervention group.

DETAILED DESCRIPTION:
The purpose of this pilot study is to determine whether augmenting an injury prevention program (IPP) with individualized video, verbal, and tactile feedback is more effective than implementation of an IPP with general education alone in female collegiate lacrosse players.

The investigators will recruit a purposive sample of 20 women from the SDSU Women's NCAA Division I Lacrosse team to conduct a quasi-experimental pilot study. To ensure adequate exposure to injury risk during matches, players who regularly participate in matches will be identified by athletics staff and offered the opportunity to participate in the study. Athletes who participate will be assigned (non-random) to one of two groups, control (education only) or education with individualized feedback, which will be balanced based on position, playing time, and history of injury.

All athletes and medical staff for the women's lacrosse team will attend a pre-season educational program focused on the purpose and benefits of IPPs, the importance of adherence to the IPP, and proper form when performing movements in the IPP to maximize injury prevention benefits. The program includes demonstration and practice of proper form, identification and correction of common errors and compensations. Videos and written documentation of the program will be shared with athletes, coaches and medical staff for reference. The athletes and staff will be encouraged to provide feedback to one another, to detect and correct errors and compensations, and help each other perform the program most optimally. This education program is scheduled to be implemented with all women's lacrosse athletes, regardless of whether the athletes participate in this research, as a joint effort between the principal investigator of the study and athletics staff, to address injury prevention for these athletes. The 10 participants assigned to the education with individualized feedback group will receive 3 additional sessions in which they receive individualized feedback on their movement when performing the IPP with one of 6 DPT students (supervised by PI Gombatto, licensed Physical Therapist). Individual feedback sessions will be 45-60 minutes and consist of a video review of athlete performance of the IPP, real-time feedback using a mirror, a combination of verbal and tactile feedback, and integration of peer feedback with a partner who is also receiving individualized feedback.

All participants (N=20) will complete pre-intervention (pre-season) and post-intervention (post-season) testing including a 3D biomechanics analysis, anthropometric and body composition measures, and questionnaires to identify other known risk factors for injury. The 3D biomechanical analysis will include an evaluation of lower extremity movement and forces with the Drop Vertical Jump (DVJ) and three directions of the Star Excursion Balance Test (SEBT). Injury history and incidence of injuries during the 2022 and 2023 season will be gathered from the athlete's electronic health records and via athlete self-report. Participant questionnaires will include questions about position, footwear, orthotic use, and taping. Adherence surveys will be administered weekly (15-16 weeks) via personalized text links or phone call (for non-responders) to record how often athletes are engaging in the IPP, self-correction, and peer feedback.

The primary outcomes of this study will be biomechanical risk factors associated with knee injury, including dynamic knee valgus during the DVJ and asymmetry in lower extremity reach distance during the SEBT. Secondary outcomes will include lower extremity injuries during the Spring 2023 season, examined between treatment groups, and for all participants between the Spring 2022 and Spring 2023 seasons. The primary outcome was selected because the intervention is proposed to change movements that place athletes at risk for injury, and injury is the secondary outcome because reduced injuries are the intended effect of the IPP but the sample size may not be sufficient to measure change in injuries during a single season with this pilot study.

Summary statistics for all outcomes will be examined for each treatment group. Analysis of variance (ANOVA) will be conducted to determine whether change in biomechanical risk factors is different between athletes in the education vs. education with individualized feedback groups (group x time interaction effect). Fisher's exact test will be used to test for differences in incidence of injury between groups. Number of lower extremity injuries across all participants will be quantitatively compared for the 2022 vs. 2023 season. Effect sizes (Cohen's d) will be calculated for each outcome. A power analysis will be performed to determine the number of subjects needed to detect significant effects in a larger sample.

ELIGIBILITY:
Inclusion Criteria:

* Athletes currently a member of the SDSU Women's NCAA Division I Lacrosse team.
* Athletes who regularly participate in games as identified by athletics staff.

Exclusion Criteria:

* Athletes deemed ineligible to participate in their sport by the team's medical staff because of an injury.
* Athletes who do not regularly participate in games throughout the season.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-01-06 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Initial Contact Knee Valgus During Drop Vertical Jump | Change from Baseline to Post-Season Biomechanics Assessment (15-16 weeks later)
  Knee Valgus Angle at Initial Contact
Maximum Knee Valgus during Drop Vertical Jump | Change from Baseline to Post-Season Biomechanics Assessment (15-16 weeks later)
  Maximum Knee Valgus Angle During Landing
Initial Contact Knee Flexion during Drop Vertical Jump | Change from Baseline to Post-Season Biomechanics Assessment (15-16 weeks later)
  Knee Flexion Angle at Initial Contact
Maximum Knee Flexion during Drop Vertical Jump | Change from Baseline to Post-Season Biomechanics Assessment (15-16 weeks later)
  Maximum Knee Flexion Angle During Landing
Force Asymmetry during Drop Vertical Jump | Change from Baseline to Post-Season Biomechanics Assessment (15-16 weeks later)
  Difference between left and right Maximum Vertical Ground Reaction Force During Landing
Reach Distance During Anterior Direction of the Star Excursion Balance Test | Change from Baseline to Post-Season Biomechanics Assessment (15-16 weeks later)
  Left and right maximum reach distances, normalized to leg length
Reach Distance During Posterior-Medial Direction of the Star Excursion Balance Test | Change from Baseline to Post-Season Biomechanics Assessment (15-16 weeks later)
  Left and right maximum reach distances, normalized to leg length
Reach Distance During Posterior-Lateral Direction of the Star Excursion Balance Test | Change from Baseline to Post-Season Biomechanics Assessment (15-16 weeks later)
  Left and right maximum reach distances, normalized to leg length
Composite Reach Distance During the Star Excursion Balance Test | Change from Baseline to Post-Season Biomechanics Assessment (15-16 weeks later)
  Average normalized maximum reach distances across the anterior, posterior-medial, and posterior-lateral directions (right and left calculated separately).
Reach Distance Asymmetry During Anterior Direction of the Star Excursion Balance Test | Change from Baseline to Post-Season Biomechanics Assessment (15-16 weeks later)
  Difference between left and right maximum reach distances (in centimeters)
Reach Distance Asymmetry During Posterior-Medial Direction of the Star Excursion Balance Test | Change from Baseline to Post-Season Biomechanics Assessment (15-16 weeks later)
  Difference between left and right maximum reach distances (in centimeters)
Reach Distance Asymmetry During Posterior-Lateral Direction of the Star Excursion Balance Test | Change from Baseline to Post-Season Biomechanics Assessment (15-16 weeks later)
  Difference between left and right maximum reach distances (in centimeters)

SECONDARY OUTCOMES:
Frequency of Injuries in Current Season | up to 16 weeks
  Number of lower extremity injuries documented in the athlete's Electronic Health Record during the Spring 2023 Season.
Frequency of Injuries in Prior Season | up to 12 months
  Number of lower extremity injuries documented in the athlete's Electronic Health Record during the prior Spring 2022 season.

OTHER OUTCOMES:
Participant Information | Baseline
  Participant date of birth, age, sex at birth, limb dominance, primary position, playing time, glasses/contacts, footwear, brace, orthotic or taping use, current medication, and injury history.
Height | Baseline
  Measured height in inches
Weight | Baseline
  Measured weight in pounds
Leg Length | Baseline
  Measured right and left leg length in centimeters
Weekly Athlete Adherence Questionnaire Adherence to Components | Weekly throughout the study (15-16 weeks)
  Self-reported adherence to the components of the injury prevention program. "Did you do all of the activities?" (Yes/No)
Weekly Athlete Adherence Questionnaire Adherence to Instructions | Weekly throughout the study (15-16 weeks)
  Self-reported adherence to the instructions for the injury prevention program. "Were you able to complete the movements in the way that you were instructed to?" (Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Sara P Gombatto, PT, PhD, Principal Investigator — San Diego State University
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
This is a pilot study. We do not plan to make individual participant data available to other researchers.